CLINICAL TRIAL: NCT01398592
Title: Cross-over Study to Assess the Difference in Fasting Plasma Glucose (FPG) Between Vildagliptin (Galvus®/Eucreas®) and Sitagliptin (Januvia®/Janumet®) After Two Weeks
Brief Title: Vildagliptin Versus Sitagliptin - Differences in Fasting Plasma Glucose Lowering Efficacy
Acronym: FPG-VISIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLMF237ADE02; 2011-000518-21 (EudraCT Number)
Record Dates: First submitted 2011-07-15; First posted 2011-07-20 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Diabetes mellitus Type two; T2DM; vildagliptin; sitagliptin; FPG; DPP-4
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; Sitagliptin Phosphate

ARMS (2):
- Vildagliptin (Experimental): Experimental
  Interventions: Drug: Vildagliptin
- Sitagliptin (Active Comparator): Active comparator (drug)
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Vildagliptin — 50mg vildagliptin bid
  Arms: Vildagliptin
Drug: Sitagliptin — 100mg sitagliptin po qd
  Arms: Sitagliptin

SUMMARY:
This study is designed to assess the potential difference in Fasting Plasma Glucose (FPG) lowering efficacy between the two DPP-4 inhibitors vildagliptin and sitagliptin, both after a two weeks treatment on top of metformin.

ELIGIBILITY:
Inclusion Criteria:

Patients with type 2 diabetes 18 to 85 years Metformin monotherapy > 4 weeks HbA1c 6.5 - 9.5%

Exclusion Criteria:

FPG > 270 mg/dl Use of other antidiabetic drugs than metformin major cardiovascular event in the last 6 months (MI, stroke…)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
demonstrate that the FPG after 14 days of treatment with Vildagliptin is superior to the FPG after 14 days of treatment with Sitagliptin | 14 days
  Fasting Plasma Glucose measured on day 14.

SECONDARY OUTCOMES:
To assess the difference in FPG between vildagliptin and sitagliptin in patients with type 2 diabetes mellitus on concomitant treatment with metformin | 14 days
  Fasting Plasma Glucose on day 14 analyzed descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Rüdiger Göke, MD, Principal Investigator — Kirchhain
Locations (12):
- Germany (12):
  - Novartis Investigative Site, Bad Oeynhausen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Celle
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Kirchhain
  - Novartis Investigative Site, Lehrte
  - Novartis Investigative Site, Mülheim
  - Novartis Investigative Site, Oberhausen
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Stuttgart

REFERENCES:
- [Derived] Goke R, Eschenbach P, Dutting ED. Efficacy of vildagliptin and sitagliptin in lowering fasting plasma glucose: Results of a randomized controlled trial. Diabetes Metab. 2015 Jun;41(3):244-7. doi: 10.1016/j.diabet.2014.07.004. Epub 2014 Nov 11. PMID 25457473